CLINICAL TRIAL: NCT05742386
Title: Evaluating the Impact of Optimizing the Use of HPV Vaccine Standing Orders in Primary Care Clinics
Brief Title: Impact of Standing Orders Optimization
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IMPACTP1SO; 5P01CA250989-02 (NIH)
Record Dates: First submitted 2023-02-13; First posted 2023-02-24 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Human Papilloma Virus
Keywords: Human Papilloma Virus; Pediatric medicine; Primary care; Standing orders; Vaccination

STUDY DESIGN:
Intervention Model Description: Cluster randomized design in which clinics will be randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPV vaccine communication training (Experimental): Staff in clinics randomized to this arm will receive an intervention called Announcement Approach Training (AAT). This training is designed to improve communication about HPV vaccination.
  Interventions: Behavioral: Communication training
- HPV vaccine communication training and standing orders optimization (Experimental): Staff in clinics randomized to this arm will receive the AAT and conduct a set of activities to optimize use of HPV vaccine standing orders.
  Interventions: Behavioral: Communication training enhanced with standing orders optimization

INTERVENTIONS:
Behavioral: Communication training — Clinics will host an AAT workshop. A trained facilitator will use a standard script and slides to deliver workshop in-person or over Zoom; clinical staff who are unavailable will take the workshop later on their own.
  Arms: HPV vaccine communication training
Behavioral: Communication training enhanced with standing orders optimization — Clinics will host an AAT workshop, as in the other trial arm.
  Clinic representatives will attend working meetings on putting HPV vaccine standing orders into clinic workflow. Clinics will then orient their staff to the standing orders. Finally, clinic representatives will discuss their use of standing orders in a learning collaborative.
  Arms: HPV vaccine communication training and standing orders optimization

SUMMARY:
This trial will look at the impact of optimizing human papillomavirus (HPV) vaccine standing orders. The research team will work with primary care clinics. Some clinics will receive communication training. Other clinics will receive the same training and tools for increasing the use of their standing orders.

DETAILED DESCRIPTION:
The researchers will conduct a cluster randomized clinical trial. The trial will look at the impact of optimizing HPV vaccine standing orders. The recruitment goal for the trial is 34 clinics in healthcare systems, including 9 rural-serving clinics. The researchers will randomize clinics using simple randomization (1:1). Some clinics will receive a communication training. Other clinics will receive a communication training and tools for optimizing the use of their standing orders. The researchers will use medical record data to compare changes in HPV vaccination among children ages 9-12. Clinics will be followed for 24 months. The researchers will also use survey data to compare HPV vaccine communication and implementation of standing orders among clinical staff. The study will engage clinical staff. Researchers will not have direct contact with children or their families.

ELIGIBILITY:
This trial will enroll clinics and intervene with clinical staff. We will use vaccination data from children and survey data from clinical staff to evaluate intervention effectiveness. We will not enroll children or interact with them directly.

Inclusion Criteria

Clinics are eligible if they:

* provide HPV vaccine to children ages 9-12
* have standing orders for HPV vaccination approved but not routinely used or be willing to adopt them prior to the start of the trial
* have rates of HPV vaccination (≥1 dose) below 72%, boys and girls combined

Children's medical records will be eligible to be included in the dataset if children:

* are between the ages of 9-12 years at baseline
* are attributed to a participating clinic at 12- or 24-month follow-up

Clinical staff's survey data will be eligible to be included in the dataset if clinical staff complete the follow-up survey.

Exclusion Criteria

Clinics are excluded if they:

* do not provide HPV vaccine to children ages 9-12
* do not have standing orders for HPV vaccination or are not willing to adopt them prior to the start of the trial
* have rates of HPV vaccination (≥1 dose) above 72%, boys and girls combined
* have hosted an AAT workshop in the previous 3 years or are part of current HPV vaccine communication trainings
* have quality improvement efforts to change HPV vaccine standing orders during the trial

Children's medical records will not be eligible to be included in the dataset if children:

* are not between the ages of 9-12 years at baseline
* are not attributed to a participating clinic at 12- or 24-month follow-up
* are receiving hospice/palliative care, are pregnant, or have a history of HPV vaccine contraindications

Clinical staff's survey data will be not eligible to be included in the dataset if clinical staff do not complete the follow-up survey.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
HPV vaccination (≥1 dose), 9-12 year olds | from baseline to 12 months
  Proportion of unvaccinated children who initiate the HPV vaccine series between baseline and 12-month follow-up, among those who were ages 9-12 at baseline.

SECONDARY OUTCOMES:
HPV vaccination (≥1 dose), 9-12 year olds | from 13 months to 24 months
  Proportion of unvaccinated children who initiate the HPV vaccine series between 13- and 24-month follow-up, among those who were ages 9-12 at 13 months.
HPV vaccination (≥2 doses), 9-12 year olds | from baseline to 12 months
  Proportion of unvaccinated children who complete the HPV vaccine series between baseline and 12-month follow-up, among those who were ages 9-12 at baseline.
HPV vaccination (≥2 doses), 9-12 year olds | from 13 months to 24 months
  Proportion of unvaccinated children who complete the HPV vaccine series between 13- and 24-month follow-up, among those who were ages 9-12 at 13 months.
Standing orders attitude rating | up to 6 months
  Positive attitude toward using HPV vaccine standing orders will be measured by one item on the survey, taken by clinical staff two months after attending the AAT. The range for this measure will be 1 to 5, with higher values indicating more positive attitudes.
Standing orders norms rating | up to 6 months
  Norms in favor of using HPV vaccine standing orders will be measured by one item on the survey, taken by clinical staff two months after attending the AAT. The range for this measure will be 1 to 5, with higher values indicating more supportive norms.
Standing orders self-efficacy rating | up to 6 months
  Confidence about using HPV vaccine standing orders will be measured by one item on the survey, taken by clinical staff two months after attending the AAT. The range for this measure will be 1 to 5, with higher values indicating higher confidence.
Standing orders adoption rating | up to 6 months
  Adoption of HPV vaccine standing orders will be measured by one item on the survey, taken by clinical staff two months after attending the AAT. The range for this measure will be 1 to 5, with higher values indicating greater adoption.
Standing orders acceptability rating | up to 6 months
  Acceptability of HPV vaccine standing orders will be measured by one item on the survey, taken by clinical staff two months after attending the AAT. The range for this measure will be 1 to 5, with higher values indicating higher acceptability.
Standing orders appropriateness rating | up to 6 months
  Appropriateness of HPV vaccine standing orders will be measured by one item on the survey, taken by clinical staff two months after attending the AAT. The range for this measure will be 1 to 5, with higher values indicating greater appropriateness.
Standing orders role rating | up to 6 months
  Understanding of role under HPV vaccine standing orders will be measured by one item on the survey, taken by clinical staff two months after attending the AAT. The range for this measure will be 1 to 5, with higher values indicating better understanding of role.
Standing orders feasibility rating | up to 6 months
  Feasibility of HPV vaccine standing orders will be measured by one item on the survey, taken by clinical staff two months after attending the AAT. The range for this measure will be 1 to 5, with higher values indicating greater feasibility.
Standing orders sustainability rating | up to 6 months
  Sustainability of HPV vaccine standing orders will be measured by one item on the survey, taken by clinical staff two months after attending the AAT. The range for this measure will be 1 to 5, with higher values indicating greater sustainability.
Estimated time spent on recommendations | up to 6 months
  Time spent on HPV vaccine recommendations will be measured by one item on the survey, taken by clinical staff two months after attending the AAT. The range for this measure will be 0-99 minutes, with higher values indicating more time spent.
Estimated recommendation frequency, 9-10 year olds | up to 6 months
  Frequency of recommending HPV vaccine for children ages 9 or 10 will be measured by one item on the survey, taken by clinical staff two months after attending the AAT. The range for this measure will be 1 to 5, with higher values indicating more frequent recommendations.
Estimated recommendation frequency, 11-12 year olds | up to 6 months
  Frequency of recommending HPV vaccine for children ages 11 or 12 will be measured by one item on the survey, taken by clinical staff two months after attending the AAT. The range for this measure will be 1 to 5, with higher values indicating more frequent recommendations.
Recommendation attitudes rating | up to 6 months
  Positive attitudes toward recommending HPV vaccine for ages children ages 9 or 10 years will be measured by one item on the survey, taken by clinical staff two months after attending the AAT. The range for this measure will be 1 to 5, with higher values indicating more positive recommendation attitudes.
Recommendation self-efficacy rating | up to 6 months
  Confidence in recommending HPV vaccine for children ages 9 or 10 will be measured by one item on the survey, taken by clinical staff two months after attending the AAT. The range for this measure will be 1 to 5, with higher values indicating higher recommendation confidence.
Recommendation norms rating | up to 6 months
  Norms in favor of recommending HPV vaccine for children ages 9 or 10 will be measured by one item on the survey, taken by clinical staff two months after attending the AAT. The range for this measure will be 1 to 5, with higher values indicating more supportive norms.
Recommendation intentions rating | up to 6 months
  Intentions to recommend HPV vaccine for children ages 9 or 10 will be measured by one item on the survey, taken by clinical staff two months after attending the AAT The range for this measure will be 1 to 5, with higher values indicating higher recommendation intentions.

CONTACTS AND LOCATIONS:
Overall Officials: Noel T Brewer, PhD, Principal Investigator — University of North Carolina
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-05-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT05742386/SAP_001.pdf